CLINICAL TRIAL: NCT07111624
Title: Comparison Between a New Crowding Indicator and the Perception of Healthcare Workers in the Emergency Department
Brief Title: A New Crowding Indicator in the Emergency Department
Status: Not yet recruiting | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: CAOS
Record Dates: First submitted 2025-07-23; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-05

CONDITIONS: Emergency Department; Crowding
MeSH Terms: conditions — Emergencies; Crowding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elegible population: All patients arrived in ED during the year 2024 and patientes arrived in the period of active monitoring of the perception of crowding.

SUMMARY:
Fenice has proposed a new indicator to measure the level of crowding in the ER. The aim of this study is to evaluate, in a national multicenter context, the degree of agreement between the Fenice indicator and the perception of crowding of the ER operators and to compare this agreement with that between NEDOCS and the perception of the operators.

DETAILED DESCRIPTION:
The NEDOCS (National Emergency Department OverCrowding Study) is currently the most widely used indicator in Italy to measure the level of crowding in Emergency Departments (EDs). However, despite its widespread use, it presents several critical issues. First of all, it was developed in a context very different from the current Italian one, since it was built on data collected in 2002 in 8 medium-large US university EDs. It is therefore not possible to take for granted that this indicator can accurately describe the current crowding conditions of Italian EDs. Furthermore, the factors that make up the NEDOCS are often calculated differently by the various hospital facilities, compromising the comparability of the estimates.

Fenice has proposed a new indicator to measure the level of crowding in EDs. The indicator was developed to measure one of the objective consequences of crowding in EDs, namely the increase in waiting time for patients with a problem classified as minor urgency or deferrable to triage (codes 3 and 4). In parallel, the Fenice study has shown that NEDOCS is not very sensitive to this objective consequence of crowding.

The aim of this study is to evaluate, in a national multicenter context, the degree of agreement between the Fenice indicator and the perception of crowding of the operators of the ER and to compare this agreement with that between NEDOCS and the perception of the operators.

ELIGIBILITY:
Inclusion Criteria:

Patients that are in EDs at the time of the survey

Exclusion Criteria:

Patients that are in EDs, but not at the time of the survey

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients arriving in the emergency department at the time of the survey.
Sampling Method: Non-Probability Sample
Enrollment: 828 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of variation in the ED staff perceived crowding level that is explained by the Fenice crowding score. | September 2025 - December 2025
  The outcome will be measured using the coefficient of determination (referred to as R2) of the linear model regressing the perceived level of crowding on the Fenice score.

SECONDARY OUTCOMES:
Proportion of variation in the ED staff perceived crowding level that is explained by the NEDOCS score, measured using the coefficient of determination (R2) of the linear model regressing the perceived level of crowding on the NEDOCS score. | September 2025 - December 2025

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Nattino, Study Chair — Istituto di Ricerche Farmacologiche Mario Negri IRCSS
Locations (10):
- Italy (10):
  - Spedali civili, Brescia, BS
  - IRCCS San Martino, Genova, GE
  - Ospedale Santa Maria delle Croci, Ravenna, RA
  - Ospedali riuniti di Anzio e Nettuno, Anzio, RM
  - Azienda Ospedaliera San Camillo Forlanini, Roma, RM
  - Presidio Osped. Riunito, Cirié, TO
  - AOU San Luigi Gonzaga, Orbassano, TO
  - P.O. Sant'Andrea, Vercelli, VC
  - AOU Maggiore della Carità, Novara
  - Ospedale Santa Maria delle Grazie, Pozzuoli

IPD SHARING:
Plan to Share IPD: Undecided